CLINICAL TRIAL: NCT00635115
Title: The VEPRO Trial: A Cross-Over Randomised Controlled Trial Comparing 2 Corrective Lenses for Patients With Presbyopia
Acronym: VEPRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Santéclair (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: FFSA-2005-01
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2008-03

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Device: a new generation of corrective lens for presbyopia (i.e., Varilux Panamic Orma Crizal)
- 2 (Active Comparator)
  Interventions: Device: an old generation of corrective lens for presbyopia (i.e., Varilux Comfort Orma Crizal)

INTERVENTIONS:
Device: a new generation of corrective lens for presbyopia (i.e., Varilux Panamic Orma Crizal)
  Other Names: VARILUX PANAMIC ORMA CRIZAL; Essilor (R)
  Arms: 1
Device: an old generation of corrective lens for presbyopia (i.e., Varilux Comfort Orma Crizal)
  Other Names: VARILUX COMFORT ORMA CRIZAL; Essilor (R)
  Arms: 2

SUMMARY:
The VEPRO trial is a cross-over randomised controlled trial comparing 2 corrective lenses for patients with presbyopia. The aim of the study is to compare the effectiveness of two corrective lenses: an old generation (Varilux Comfort Orma Crizal) and a new generation (Varilux Panamic Orma Crizal) of corrective lenses prescribed in presbyopia.

ELIGIBILITY:
Inclusion Criteria:

* age 43 to 60 years old
* outpatients wearing corrective lenses for presbyopia, referred to an optician within the last 6 months for a change in their optical correction
* associated hyperopia or astigmatism, the required correction had to be ≤ 3 dioptres in that case
* understanding, speaking French and able to answer a questionnaire

Exclusion Criteria:

* first prescription of corrective lenses for presbyopia
* associated strabism
* associated amblyopia
* orthoptics therapy
* associated anisometropia > 1.5 dioptres
* patients treated for diabetes

Ages: 43 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2006-02; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
patient preference for a corrective lens | 8 weeks

SECONDARY OUTCOMES:
subjective measures of different areas of visual performance. | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- INSERM, U738, Paris, France ; Université Paris 7 Denis Diderot, UFR de Médecine, Paris, France ; AP-HP, Hôpital Bichat, Département d'Epidémiologie, Biostatistique et Recherche Clinique, Paris, France

REFERENCES:
- [Derived] Boutron I, Touizer C, Pitrou I, Roy C, Ravaud P. The VEPRO trial: a cross-over randomised controlled trial comparing 2 progressive lenses for patients with presbyopia. Trials. 2008 Sep 19;9:54. doi: 10.1186/1745-6215-9-54. PMID 18803826